CLINICAL TRIAL: NCT05309460
Title: Labetalol or Nifedipine for Control of Postpartum Hypertension: A Randomized Controlled Trial
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nebraska Methodist Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NebraskaMethodistHS
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Postpartum Preeclampsia; Hypertension in Pregnancy
Keywords: Nifedipine; Labetalol; Postpartum; Hypertension; Preeclampsia; Pregnancy
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Hypertension; Pre-Eclampsia | interventions — Labetalol; Nifedipine

STUDY DESIGN:
Intervention Model Description: Two arm, block randomized Arm A: Nifedipine Arm B: Labetalol
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nifedipine (Active Comparator): Patients randomized to Nifedipine will be started on Nifedipine XR 30mg BID. Escalation in therapy to be determined by primary provider. Maximum dose of Nifedipine is 120mg daily. All patients will be monitored for signs and symptoms of hypotension or medication side effect- severe HA, orthostasis, syncope.
  Interventions: Drug: NIFEdipine ER
- Labetalol (Active Comparator): Patients randomized to Labetalol will be started on 200mg TID. Escalation in therapy to be determined by primary provider. Maximum dose is 2400mg in a day. All patients will be monitored for signs and symptoms of hypotension or medication side effect- orthostasis, syncope, bradycardia.
  Interventions: Drug: Labetalol Oral Tablet

INTERVENTIONS:
Drug: Labetalol Oral Tablet — See Labetalol arm.
  Other Names: Normodyne; Trandate
  Arms: Labetalol
Drug: NIFEdipine ER — See Nifedipine arm.
  Other Names: Procardia XL
  Arms: Nifedipine

SUMMARY:
Randomized trial comparing risk of hospital readmission and hypertensive complications between patients managed on Labetalol compared to Nifedipine.

DETAILED DESCRIPTION:
Enrollment:

Patients will be identified daily using an EMR screening tool. Those that meet inclusion criteria will then be approached by the investigators or research RN for enrollment. Patients consenting to be involved in the study will then be randomly assigned to the nifedipine or labetalol arms of the study. Block randomization will be performed in blocks of 50 with goal of 600 total patients (300 in each arm).

Treatment Protocols

Nifedipine Study Arm:

Patients randomized to Nifedipine will be started on Nifedipine XR 30mg BID. Escalation in therapy to be determined by primary provider. Maximum dose of Nifedipine is 120mg daily. All patients will be monitored for signs and symptoms of hypotension or medication side effect- severe HA, orthostasis, syncope. Patients with further hypertension will then be started on Labetalol as a second agent at 200mg TID and escalated as needed with the goal of being normotensive for at least 12 hours before discharge. Patients will not be kept hospitalized for purposes of the study.

Labetalol Study Arm:

Patients randomized to Labetalol will be started on 200mg TID. Escalation in therapy to be determined by primary provider. Maximum dose is 2400mg in a day. All patients will be monitored for signs and symptoms of hypotension or medication side effect- orthostasis, syncope, bradycardia. Patient's that reach 800mg TID or cannot escalate therapy due to bradycardia will then be started on Nifedipine 30mg BID and escalated as needed with the goal of normotension for at least 12 hours before discharge. Patients will not be kept hospitalized for purposes of the study.

All Patients:

Outpatient follow up to be dictated by the discharging provider. Patients will be called at 6 months to determine if they were readmitted and their MRN will be used to query the EMR for readmission or ER evaluation.

Power Calculation Anticipated incidence in Nifedipine arm is 1%. Pilot study indicated a readmission risk of 0.2% in patients discharge normotensive on nifedipine. We anticipate this will be higher as some patients will likely be discharged with HTN. Anticipated incidence in the Labetalol arm is 7%. This number was based on a 5.8% risk of readmission in the normotensive group and 12.6% in the hypertensive group. As with the nifedipine arm, we anticipate there will be some patients discharged hypertensive increasing this risk above that of patients discharged normotensive.

With alpha set at 0.05 and power of 80%, we anticipate we will need at least 332 total patients, 166 in each arm. The original pilot data included patients with both physician identified hypertensive disease as well as those patients only identified by the EMR screening tool. Those patients identified by the screening tool had an increased risk of readmission compared to the overall population based risk of readmission (3.6% vs 1%). Their risk is lower than those patients identified by their provider 5.2%. Our plan is to enroll 600 patients, 300 in each arm as some patients will require multiple medications and due to the dilution of including a lower risk group we feel the initial power calculation does not take these factors into account. All data will be analyzed by intention to treat and crossover between groups for side effects or primary physician change in management will be reported/monitored.

Data Safety Monitoring Data will be reviewed q 6 months for statistical significance once at least 100 patients have been enrolled in each arm. If the effect is statistically significant to a p of 0.05 the study will be terminated for safety reasons. The DSMB will also monitor patient crossover and medication side effects as part of their evaluation. Data safety monitoring board will be comprised of 2 maternal fetal medicine physicians, 1 general obstetrician and the study research RN. Data will be analyzed as each block in the randomization is completed.

ELIGIBILITY:
Inclusion Criteria:

Any patient admitted for delivery by cesarean or vaginal delivery at 24 weeks gestation or greater with hypertension(HTN). Hypertension will be defined during the study as either a systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg on two occasions at least 4 hours apart. This definition is consistent with the ACOG definition for pregnancy related HTN. Following enrollment, treatment will be escalated at discretion of primary provider with the goal of normotension.

Exclusion Criteria:

History of moderate persistent asthma, coronary artery disease, heart failure, AV heart block, pulmonary edema

* Contraindication to either Nifedipine or Labetalol
* HR <60 or >110
* Native language other than English or Spanish

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Readmission | 6 months
  Patients will be monitored following delivery for readmission to the hospital. To improve patient capture, all patients will be called at 6 months to identify complications or if hospital admission occured in the 6 months following delivery

SECONDARY OUTCOMES:
Medication failure | Any time during the 6 months following delivery
  Need for additional antihypertensive medication
Medication change or discontinuation | Any time during the 6 months following delivery
  Need to change medication or discontinue medication due to side effects or complications of medication.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Lovgren, MD, Principal Investigator — Nebraska Methodist Health System
Locations (1):
- Nebraska Methodist Women's Hospital, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Yes, deidentified data will be shared on a case by case basis.
Supporting Information: Study Protocol
Time Frame: On completion of study for 12 months.
Access Criteria: TBD by primary author.

REFERENCES:
- [Background] Lovgren T, Connealy B, Yao R, Dahlke JD. Postpartum management of hypertension and effect on readmission rates. Am J Obstet Gynecol MFM. 2022 Jan;4(1):100517. doi: 10.1016/j.ajogmf.2021.100517. Epub 2021 Oct 30. PMID 34757235
- [Background] Lovgren T, Connealy B, Yao R, D Dahlke J. Postpartum medical management of hypertension and risk of readmission for hypertensive complications. J Hypertens. 2023 Feb 1;41(2):351-355. doi: 10.1097/HJH.0000000000003340. Epub 2022 Dec 13. PMID 36511111